CLINICAL TRIAL: NCT05683561
Title: A Randomized, Double-blind, Positive-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of SCTV01E (A COVID-19 Alpha/Beta/Delta/Omicron Variants S-Trimer Vaccine) in Healthy People
Brief Title: A Phase III Clinical Trial to Evaluate the Efficacy and Safety of SCTV01E in Healthy People
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SCTV01E-MRCT-1
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: COVID-19 SARS-CoV-2 Infection
MeSH Terms: interventions — sinovac COVID-19 vaccine; SCTV01C vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CoronaVac (Active Comparator): one dose of CoronaVac on D0
  Interventions: Biological: CoronaVac
- SCTV01E (Experimental): one dose of SCTV01E on D0
  Interventions: Biological: SCTV01E

INTERVENTIONS:
Biological: CoronaVac — D0; intramuscular injection
  Arms: CoronaVac
Biological: SCTV01E — D0; intramuscular injection
  Arms: SCTV01E

SUMMARY:
The objective of this study is to evaluate the effectiveness of SCTV01E in healthy people

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo-controlled Phase III study. It will evaluate the protective effectiveness and safety of SCTV01E against COVID-19 in participants who were previously received primary series or booster dose of COVID-19 vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years old when signing ICF (the specific age range depends on the authorized age range by local regulatory authority);
2. Participants who were vaccinated with primary series COVID-19 vaccine and/or received booster vaccination, and the last dose of COVID-19 vaccine was received more than 3 months;
3. The participant and/or his/her legal guardian and/or his entrusted person can sign written ICF, and can fully understand the trial procedure, the risk of participating in the trial, and other interventions that can be selected if they do not participate in the trial;
4. The baseline SARS-CoV-2 anti-Spike IgG will be measured at the screening period and an upper IgG limit may be used to screen the participants. It is aimed to recruit participants who are susceptible to SARS-CoV-2 infection. The participant with the IgG level higher than the limit may be excluded from the study. The IgG limit will be determined based on the average level of IgG in a region, and may not be applied if the incidence rate of COVID-19 is low;
5. The participant and/or his/her legal guardian and/or his entrusted person have the ability to read, understand, and fill in record cards;
6. Healthy participants or participants with pre-existing medical conditions who are in stable condition. The "pre-existing medical conditions" include but not limited to hypertension, diabetes, Chronic cholecystitis and cholelithiasis, chronic gastritis that meet the described criteria. A stable medical condition is defined as disease not requiring significant change in therapy or no need for hospitalization as a consequence of worsening disease state for at least 3 months prior to enrollment;
7. Fertile men and women of childbearing potential voluntarily agree to take effective contraceptive measures from signing ICF to 6 months after the last dose of study vaccination; the pregnancy test results of women of childbearing potential are negative on screening.

Exclusion Criteria:

1. A positive result of nucleic acid test or rapid antigen test for SARS-CoV-2 during the screening period;
2. Known history of SARS-CoV-2 infection in past 6 months before the study vaccination;
3. Presence of fever within 3 days before the study vaccination;
4. A history of severe allergic reactions to any vaccines or drugs, such as severe skin eczema, dyspnea, laryngeal edema, and angioneurotic edema;
5. A medical or family history of seizure, epilepsy, encephalopathy and psychosis;
6. Immunocompromised patients suffering from immunodeficiency diseases, important organ diseases, immune diseases (including Guillain-Barre Syndrome [GBS], systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy caused by any circumstances, and other immune diseases that may have an impact on immune response in the investigator's opinion), etc.;
7. Long-term use of immunosuppressant therapy or immunomodulatory drugs for >14 days within the six months prior to enrollment. Whereas short-term (≤14 days) use of oral, inhaled and topical steroids are allowed;
8. Patients on antituberculosis therapy;
9. Presence of severe or uncontrollable cardiovascular diseases, or severe or uncontrollable disorders related to endocrine system, blood and lymphatic system, liver and kidney, respiratory system, metabolic and skeletal systems, or malignancies (skin basal cell carcinoma and carcinoma in-situ of cervix are exceptions and will not be excluded), such as severe heart failure, severe pulmonary heart disease, unstable angina, liver failure, or uremia;
10. Contraindications for intramuscular injection or intravenous blood sampling, including thrombocytopenia and other blood coagulation disorders;
11. Participants who received any immunoglobulin or blood products in the previous 3 months before enrollment, or plan to receive similar products during the study;
12. Participants who received other investigational drugs within 30 days before the study vaccination or who intend to participate in another clinical study at any time during the conduct of this study;
13. Participants who have acute illness, such as acute onset of chronic heart failure, acute sore throat, hypertensive encephalopathy, acute pneumonia, acute renal insufficiency, acute cholecystitis;
14. Participants vaccinated with influenza vaccine within 14 days or with other vaccines within 28 days before the study vaccination;
15. Those who donated blood or had blood loss (≥450 mL) within 3 months before the vaccination or plan to donate blood during the study period;
16. Those who are pregnant or breast-feeding or plan to be pregnant during the study period;
17. Those who plan to donate ovum or sperms during the study period;
18. Those who cannot follow the trial procedures, or cannot cooperate to complete the study due to planned relocation or long-term outing;
19. Those unsuitable for participating in the clinical trial as determined by the investigator because of other abnormalities that are likely to confuse the study results, or non-conformance with the maximal benefits of the participants;
20. Those who are tested positive for HIV in terms of serology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2023-01-25 (Estimated); Primary Completion 2023-08-25 (Estimated); Study Completion 2024-08-25 (Estimated)

PRIMARY OUTCOMES:
Cases of the first occurrence of symptomatic COVID-19 of any severity starting 14 days (≥15 days) after the study vaccination | From Day 15 to Day 365
  To evalute the efficacy of SCTV01E

SECONDARY OUTCOMES:
Cases of the first occurrence of symptomatic COVID-19 of any severity starting 7 days (≥8 days) after the study vaccination. | From Day 8 to Day 365
  To evalute the efficacy of SCTV01E
Cases of the first occurrence of moderate and above COVID-19, severe and above COVID-19, hospitalization due to COVID-19, and death due to COVID-19, respectively, starting 7 days (≥8 days) after the study vaccination | From Day 8 to Day 365
  To evalute the efficacy of SCTV01E
Cases of the first occurrence of moderate and above COVID-19, severe and above COVID-19, hospitalization due to COVID-19, and death due to COVID-19, respectively, starting 14 days (≥15 days) after the study vaccination. | From Day 15 to Day 365
  To evalute the efficacy of SCTV01E
Cases of the first occurrence of symptomatic COVID-19 of any severity caused by SARS-CoV-2 variants and subvariants starting 7 days (≥8 days) after the study vaccination. | From Day 8 to Day 365
  To evalute the efficacy of SCTV01E
Cases of the first occurrence of symptomatic COVID-19 of any severity caused by SARS-CoV-2 variants and subvariants starting 14 days (≥15 days) after the study vaccination. | From Day 15 to Day 365
  To evalute the efficacy of SCTV01E
Geometric mean titers (GMT) of neutralizing antibodies (nAb) against SARS-CoV-2 (including its variants and subvariants) on D28. | From Day 0 to Day 28
  To evalute the immunogenicity of SCTV01E
Incidence and severity of solicited AEs of SCTV01E from D0 to D7 | From Day 0 to Day 7
  To evalute the safety of SCTV01E
Incidence and severity of unsolicited AEs of SCTV01E from D0 to D28. | From Day 0 to Day 28
  To evalute the safety of SCTV01E
Incidence and severity of SAEs and AESIs. | From Day 0 to Day 365
  To evalute the safety of SCTV01E

CONTACTS AND LOCATIONS:
Overall Officials: Yu Sun, Study Chair — Sinocelltech Ltd.